CLINICAL TRIAL: NCT04330495
Title: Randomized, Controlled, Double-blind Clinical Trial Comparing the Efficacy and Safety of Chemoprophylaxis With Hydroxychloroquine in Patients Under Biological Treatment and / or JAK Inhibitors in the Prevention of SARS-CoV-2 Infection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: * Care pressures on the investigator team during the COVID-19 pandemic.
  * Subsequent appearance of scientific evidence on the lack of efficacy of hydroxychloroquine in the treatment or prophylaxis of COVID-19 infection.
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EnCOVID-HidroxiCLOROQUINA
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: COVID 19; Immunomediated Inflammatory Disease in Treatment With Biological Agents and / or Jak Inhibitors
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testing and prophylaxis of SARS-CoV-2 (Experimental): Chemoprophylaxis with hydroxychloroquine at a dose of 200 mg twice a day for 6 months.
  Interventions: Drug: Hidroxicloroquina
- placebo (Active Comparator): Testing of SARS-CoV-2 and prescription of placebo (Hydroxychloroquine placebo) twice daily for 6 months
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Hidroxicloroquina — Chemoprophylaxis with hydroxychloroquine at a dose of 200 mg twice a day for 6 months.
  Arms: Testing and prophylaxis of SARS-CoV-2
Drug: Control group — Testing of SARS-CoV-2 and prescription of placebo (Hydroxychloroquine placebo) twice daily for 6 months
  Arms: placebo

SUMMARY:
The investigators plan to evaluate a strategy of chemoprophylaxis with hydroxyloquine (HCQ) against COVID-19 infection in patients diagnosed with an immunomediated inflammatory disease who are following a treatment with biological agents and / or Jak inhibitors. The strategy will be carried out through a randomised double blind, placebo-controlled clinical trial and will assess comparative rates of infection (prevalence, incidence), severity including mortality, impact on clínical course of the primary diseases and toxicity. Such evaluation will require prospective surveillance to assess the different end-points.

Drug interventions in this protocol will follow the Spanish law about off-label use of medicines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the requirements of the New Coronavirus Infection Diagnosis (Acute respiratory infection symptoms or acute cough alone and positive PCR)
2. Aged ≥18 and < 75 years male or female;
3. In women of childbearing potential, negative pregnancy test and commitment to use contraceptive method throughout the study.
4. Willing to take study medication
5. Willing to comply with all study procedures,
6. Diagnosis of IBD disease, rheumatoid arthritis, seronegative spondyloarthritis or psoriasis for more than 6 months.
7. Be on stable treatment with biological agents, for a minimum period of 6 months, including treatment with Infliximab, etanercept, adalimumab, certolizumab, golimumab, rituximab, abatacept, tocilizumab, sarilumab, secukinumab, vedolizumab, natalizumab, ustekinumab, tofacit
8. Able to provide oral and written informed consent

Exclusion Criteria

1. Previous infection with SARS-CoV-2.
2. Current treatment with hydroxychloroquine / chloroquine.
3. Previous or current treatment with tamoxifen or raloxifene.
4. Previous eye disease, especially maculopathy.
5. Known heart failure grade III-IV of the classification of the New York Heart Association).
6. Any type of cancer (except basal cell) in the last 5 years.
7. Pregnancy.
8. Refusal to give informed consent.
9. Evidence of any other unstable or clinically significant unstable, clinically significant, immunological, endocrine, hematologic, gastrointestinal, neurological, neoplastic, or psychiatric illness.
10. Instability or mental incompetence, so that the validity of the informed consent or the ability to complete the study is uncertain.
11. Positive antibodies to the human immunodeficiency virus.
12. Data on decompensated liver disease:

to. Aspartate aminotransferase (AST) and / or ALT> 10 x upper limit of normal (LSN).

b. Total bilirubin> 25 μmol / l (1.5 mg / dl). c. International normalized index> 1.4. d. Platelet count <100,000 / mm3. 17. Serum creatinine levels> 135 μmol / l (> 1.53 mg / dl) in men and> 110 μmol / l (> 24 mg / dl) in women.

18.Significant kidney disease, including nephrotic syndrome, chronic kidney disease (patients with markers of liver injury or estimated glomerular filtration rate [eGFR] of less than 60 ml / min / 1.73 m2). If an abnormal value is obtained at the first screening visit, the measurement of eGFR may be repeated before randomization within the following time frame: minimum 4 weeks after the initial test and maximum 2 weeks before the planned randomization. Repeated abnormal eGFR (less than 60 ml / min / 1.73 m2) leads to exclusion from the study.Pregnant or lactating women; 19. Inability to consent and/or comply with study protocol; 20. Individuals with known hypersensitivity to the study drugs. 21. Any contraindications as per the Data Sheet of or Hydroxychloroquine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-06 (Estimated); Primary Completion 2020-11-06 (Estimated); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Incidence rate of new COVID-19 cases in both arms | From day 14 after start of treatment up to the end of follow-up: week 27
  number of new cases divided by number of persons-time at risk
Prevalence of COVID-19 cases in both arms | 27 weeks after the beginning of the study
  percentage of cases of COVID 19
Mortality rate secondary to COVID-19 cases in both groups | 27 weeks after the beginning of the study
  Case fatality rate (CFR): the proportion of diagnosed cases of COVID 19 that lead to death
Intensive Care Unit (CU) admission rate secondary to COVID-19 cases in both groups | 27 weeks after the beginning of the study
  percentage of patients who need admission in an ICU due to COVID 19 infection

SECONDARY OUTCOMES:
Adverse events | 12 weeks after the start of treatment
  Presence and type of adverse events at this point.
Adverse events | 27 weeks after the beginning of the study
  Proportion of participants that drop out of study

IPD SHARING:
Plan to Share IPD: Undecided